CLINICAL TRIAL: NCT03858530
Title: Using Ultrasound Elastography to Predict Development of Sinusoidal Obstruction Syndrome
Brief Title: Ultrasound Elastography to Predict Development of SOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow patient accrual and so Multicenter study was started that had similar aims.
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Sherwin Chan MD PhD, Physician, MD, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17110684
Record Dates: First submitted 2018-12-10; First posted 2019-02-28 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Bone Marrow Transplant Complications; Sinusoidal Obstruction Syndrome; Veno-occlusive Disease; Stem Cell Transplant Complications
Keywords: Ultrasound elastography
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All Patients Enrolled (Experimental): All patients will undergo limited abdominal US with Doppler and SWE once a week upon admission for conditioning until the patient day +30 BMT or discharge, whichever comes first. Additional ultrasounds will also be performed if SOS is suspected.
  Interventions: Diagnostic Test: Ultrasound Examination

INTERVENTIONS:
Diagnostic Test: Ultrasound Examination — Grayscale ultrasound, Doppler ultrasound, ultrasound elastography with or without ultrasound intravenous contrast will be performed.

SUMMARY:
The long-term goal of our research is to accurately identify SOS patients who would benefit from defibrotide treatment using US SWE. The overall objective of this study is to validate SWE as an early diagnostic marker for SOS. Our central hypothesis is that SWE changes will precede clinical and conventional US diagnostic criteria for SOS. Our hypothesis has been formulated on the basis of our own preliminary data. The investigators completed the first prospective cohort trial demonstrating that US SWE provides SOS diagnosis (80% sensitivity and 67% specificity) nine days earlier than current clinical criteria. SWE is widely available, has no known side effects, and is easy to learn and interpret. Our study enrolled 25 high-risk BMT patients over 18 months (five with SOS and two with severe SOS). More data is needed to determine the optimal window for testing to balance between improved test characteristics and early detection of disease. The investigators propose conducting a prospective cohort study with 80 additional patients, 12 of which will likely develop SOS (including four with severe SOS) to optimize SWE timing. This study will increase the confidence in the findings from our preliminary study and allow us to test SWE against newly published clinical criteria. The rationale for the proposed research is that, if SWE can diagnose SOS earlier than clinical criteria, then SWE can guide early initiation of SOS treatment.

DETAILED DESCRIPTION:
Hepatic sinusoidal obstructive syndrome (SOS) is a complication of blood and marrow transplant (BMT) that is associated with high morbidity and mortality. 57,000 patients in the United States and Europe undergo BMT annually, and SOS affects up to 15% of these patients. SOS pathogenesis is thought to be caused by damage to the hepatic venous endothelium due to the preparative regimen used before BMT. This damage results in obstruction of blood flow through the liver. Pathology shows collagen deposition in the sinusoids and fibrosis of venous lumens. The severity of the disease is correlated to the number and severity of the histological changes. Mild and moderate SOS can resolve with supportive treatment. Severe SOS (30% of SOS) is commonly associated with multi-organ failure and has a mortality rate of 80% despite available prophylaxis and treatment (Table 1).

SOS is most commonly defined by two clinical criteria: the modified Seattle criteria and the Baltimore criteria (Table 2). The modified Seattle criteria state that at least two of the following criteria must be present within 20 days of BMT: bilirubin > 2mg/dL; hepatomegaly and/or ascites; and/or weight gain > 5% above baseline weight. Pediatric SOS incidence in BMT is 20% and is higher compared to adults. Death or multi-organ dysfunction affects 30-60% children who develop SOS. The most common definition of severe SOS is retrospective, namely death from SOS-related causes or persistent multi-organ dysfunction at 100 days post BMT. However, the European Society for Blood and Marrow Transplantation has proposed a new prospective SOS grading scheme that will likely become standard of care since it is pediatric patient specific and it is can be performed prospectively and thus can guide treatment.

Recently, a promising drug for SOS treatment has been discovered, defibrotide, which is a DNA derivative from porcine intestine that protects and repairs endothelial cells. Prior trials showed that defibrotide decreased the incidence of multi-organ failure and death from SOS. The main caveat is that treatment must be initiated very close to the time of clinical diagnosis using the Baltimore criteria to be effective. A study showed that 31/33 (94%) patients had complete remission of their SOS when treated with defibrotide <3 days after diagnosis, whereas only 3/12 (25%) patients had complete remission when treated >3 days of diagnosis. However, universal prophylaxis is infeasible due to high drug costs ($155,000 for patient) (2016). There is a critical need for an early and effective SOS diagnostic test that can identify patients who would benefit from defibrotide treatment.

Several adult and pediatric prospective studies have evaluated the efficacy of grayscale and Doppler ultrasound (US) in diagnosing SOS and have concluded that the clinical criteria are superior to US criteria for SOS diagnosis. The main reason for this conclusion is that conventional US is able to diagnose SOS only after the clinical diagnosis. This research has resulted in multiple recent guidelines recommending US only for confirming clinical diagnoses or following disease progression and not for primary diagnosis. Ultrasound shear wave elastography (SWE) has been shown to effectively diagnose passive hepatic congestion. Fontan physiology is the best studied example. SWE values markedly increased after the Fontan operation. This surgery connects the hepatic venous circulation to the pulmonary arteries exposing the liver to increased resistance from the pulmonary circulation thereby increasing hepatic venous congestion. Additionally, the effect sizes in the Fontan studies are large compared with the effect sizes in hepatic fibrosis studies. The common thread of hepatic venous congestion between Fontan physiology and SOS physiology led us to hypothesize that SWE could be useful in SOS diagnosis. Additionally, preliminary SWE studies in adults showed that it might be useful in the setting of SOS.

Data Collection Procedures Candidates for the study will be identified by a BMT physician taking care of the patient and will be identified as a potential candidate for the study. Subjects will be approached for consent by a member of the research team prior to start of conditioning regimen. Consented subjects will have demographic, laboratory and clinical data collected from the chart at each ultrasound time point.

Ultrasound Examinations and Timeline After enrollment and within two weeks prior to starting their conditioning regimen, a limited abdominal US with Doppler measurements of the hepatic arteries, hepatic and portal veins, as well as SWE will be performed.

Subjects will be undergo US examinations based on disease course as outlined below:

1. All Patients: Patients will undergo limited abdominal US with Doppler and SWE once a week upon admission for conditioning until the patient day +30 BMT or discharge, whichever comes first.
2. Inpatient SOS: patients will undergo limited abdominal US with doppler and SWE once a week upon admission for conditioning until resolution of SOS.
3. Late Onset SOS: patients will undergo limited abdominal US with Doppler and SWE once a week upon admission for conditioning until resolution of SOS.

Clinically indicated US and SWE exams for suspicion for SOS will be included in our analysis. All imaging will be performed using General Electric Logiq E9 US machines by dedicated pediatric sonographers and interpreted by board-certified pediatric radiologists. Twelve shear wave velocity measurements will be taken 2-3 cm below the liver capsule at the mid-clavicular line in the right hepatic lobe and another 12 will be taken in the left hepatic lobe near midline avoiding areas of vasculature. By necessity, the sonographer and interpreting radiologist will not be blinded to the clinical status of the patient. US and clinical data will be collected weekly and managed using REDCap electronic data capture tools hosted at Children's Mercy Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults, ages 1 month through 21 years who are undergoing allogenic or autologous myeloablative stem cell transplant.

Exclusion Criteria:

* Any other medical or social condition that in the opinion of the investigator would make them unsuitable to participate.
* Inability to properly image patient by ultrasound (e.g. uncooperative)

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shewin Chan, MD, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shulman HM, Fisher LB, Schoch HG, Henne KW, McDonald GB. Veno-occlusive disease of the liver after marrow transplantation: histological correlates of clinical signs and symptoms. Hepatology. 1994 May;19(5):1171-81. PMID 8175139
- [Background] Mohty M, Malard F, Abecassis M, Aerts E, Alaskar AS, Aljurf M, Arat M, Bader P, Baron F, Bazarbachi A, Blaise D, Ciceri F, Corbacioglu S, Dalle JH, Dignan F, Fukuda T, Huynh A, Masszi T, Michallet M, Nagler A, NiChonghaile M, Okamoto S, Pagliuca A, Peters C, Petersen FB, Richardson PG, Ruutu T, Savani BN, Wallhult E, Yakoub-Agha I, Duarte RF, Carreras E. Revised diagnosis and severity criteria for sinusoidal obstruction syndrome/veno-occlusive disease in adult patients: a new classification from the European Society for Blood and Marrow Transplantation. Bone Marrow Transplant. 2016 Jul;51(7):906-12. doi: 10.1038/bmt.2016.130. Epub 2016 May 16. PMID 27183098
- [Background] McDonald GB, Hinds MS, Fisher LD, Schoch HG, Wolford JL, Banaji M, Hardin BJ, Shulman HM, Clift RA. Veno-occlusive disease of the liver and multiorgan failure after bone marrow transplantation: a cohort study of 355 patients. Ann Intern Med. 1993 Feb 15;118(4):255-67. doi: 10.7326/0003-4819-118-4-199302150-00003. PMID 8420443
- [Background] Jones RJ, Lee KS, Beschorner WE, Vogel VG, Grochow LB, Braine HG, Vogelsang GB, Sensenbrenner LL, Santos GW, Saral R. Venoocclusive disease of the liver following bone marrow transplantation. Transplantation. 1987 Dec;44(6):778-83. doi: 10.1097/00007890-198712000-00011. PMID 3321587
- [Background] Corbacioglu S, Cesaro S, Faraci M, Valteau-Couanet D, Gruhn B, Rovelli A, Boelens JJ, Hewitt A, Schrum J, Schulz AS, Muller I, Stein J, Wynn R, Greil J, Sykora KW, Matthes-Martin S, Fuhrer M, O'Meara A, Toporski J, Sedlacek P, Schlegel PG, Ehlert K, Fasth A, Winiarski J, Arvidson J, Mauz-Korholz C, Ozsahin H, Schrauder A, Bader P, Massaro J, D'Agostino R, Hoyle M, Iacobelli M, Debatin KM, Peters C, Dini G. Defibrotide for prophylaxis of hepatic veno-occlusive disease in paediatric haemopoietic stem-cell transplantation: an open-label, phase 3, randomised controlled trial. Lancet. 2012 Apr 7;379(9823):1301-9. doi: 10.1016/S0140-6736(11)61938-7. Epub 2012 Feb 23. PMID 22364685
- [Background] Barker CC, Butzner JD, Anderson RA, Brant R, Sauve RS. Incidence, survival and risk factors for the development of veno-occlusive disease in pediatric hematopoietic stem cell transplant recipients. Bone Marrow Transplant. 2003 Jul;32(1):79-87. doi: 10.1038/sj.bmt.1704069. PMID 12815482
- [Background] Cesaro S, Pillon M, Talenti E, Toffolutti T, Calore E, Tridello G, Strugo L, Destro R, Gazzola MV, Varotto S, Errigo G, Carli M, Zanesco L, Messina C. A prospective survey on incidence, risk factors and therapy of hepatic veno-occlusive disease in children after hematopoietic stem cell transplantation. Haematologica. 2005 Oct;90(10):1396-404. PMID 16219577
- [Background] Coppell JA, Richardson PG, Soiffer R, Martin PL, Kernan NA, Chen A, Guinan E, Vogelsang G, Krishnan A, Giralt S, Revta C, Carreau NA, Iacobelli M, Carreras E, Ruutu T, Barbui T, Antin JH, Niederwieser D. Hepatic veno-occlusive disease following stem cell transplantation: incidence, clinical course, and outcome. Biol Blood Marrow Transplant. 2010 Feb;16(2):157-68. doi: 10.1016/j.bbmt.2009.08.024. Epub 2009 Sep 18. PMID 19766729
- [Background] Richardson PG, Soiffer RJ, Antin JH, Uno H, Jin Z, Kurtzberg J, Martin PL, Steinbach G, Murray KF, Vogelsang GB, Chen AR, Krishnan A, Kernan NA, Avigan DE, Spitzer TR, Shulman HM, Di Salvo DN, Revta C, Warren D, Momtaz P, Bradwin G, Wei LJ, Iacobelli M, McDonald GB, Guinan EC. Defibrotide for the treatment of severe hepatic veno-occlusive disease and multiorgan failure after stem cell transplantation: a multicenter, randomized, dose-finding trial. Biol Blood Marrow Transplant. 2010 Jul;16(7):1005-17. doi: 10.1016/j.bbmt.2010.02.009. Epub 2010 Feb 16. PMID 20167278
- [Background] Corbacioglu S, Carreras E, Ansari M, Balduzzi A, Cesaro S, Dalle JH, Dignan F, Gibson B, Guengoer T, Gruhn B, Lankester A, Locatelli F, Pagliuca A, Peters C, Richardson PG, Schulz AS, Sedlacek P, Stein J, Sykora KW, Toporski J, Trigoso E, Vetteranta K, Wachowiak J, Wallhult E, Wynn R, Yaniv I, Yesilipek A, Mohty M, Bader P. Diagnosis and severity criteria for sinusoidal obstruction syndrome/veno-occlusive disease in pediatric patients: a new classification from the European society for blood and marrow transplantation. Bone Marrow Transplant. 2018 Feb;53(2):138-145. doi: 10.1038/bmt.2017.161. Epub 2017 Jul 31. PMID 28759025
- [Background] Corbacioglu S, Greil J, Peters C, Wulffraat N, Laws HJ, Dilloo D, Straham B, Gross-Wieltsch U, Sykora KW, Ridolfi-Luthy A, Basu O, Gruhn B, Gungor T, Mihatsch W, Schulz AS. Defibrotide in the treatment of children with veno-occlusive disease (VOD): a retrospective multicentre study demonstrates therapeutic efficacy upon early intervention. Bone Marrow Transplant. 2004 Jan;33(2):189-95. doi: 10.1038/sj.bmt.1704329. PMID 14661036
- [Background] McCarville MB, Hoffer FA, Howard SC, Goloubeva O, Kauffman WM. Hepatic veno-occlusive disease in children undergoing bone-marrow transplantation: usefulness of sonographic findings. Pediatr Radiol. 2001 Feb;31(2):102-5. doi: 10.1007/s002470000373. PMID 11214676
- [Background] Hommeyer SC, Teefey SA, Jacobson AF, Higano CS, Bianco JA, Colacurcio CJ, McDonald GB. Venocclusive disease of the liver: prospective study of US evaluation. Radiology. 1992 Sep;184(3):683-6. doi: 10.1148/radiology.184.3.1509050.
- [Background] Teefey SA, Brink JA, Borson RA, Middleton WD. Diagnosis of venoocclusive disease of the liver after bone marrow transplantation: value of duplex sonography. AJR Am J Roentgenol. 1995 Jun;164(6):1397-401. doi: 10.2214/ajr.164.6.7754881.
- [Background] Bajwa RPS, Mahadeo KM, Taragin BH, Dvorak CC, McArthur J, Jeyapalan A, Duncan CN, Tamburro R, Gehred A, Lehmann L, Richardson P, Auletta JJ, Woolfrey AE. Consensus Report by Pediatric Acute Lung Injury and Sepsis Investigators and Pediatric Blood and Marrow Transplantation Consortium Joint Working Committees: Supportive Care Guidelines for Management of Veno-Occlusive Disease in Children and Adolescents, Part 1: Focus on Investigations, Prophylaxis, and Specific Treatment. Biol Blood Marrow Transplant. 2017 Nov;23(11):1817-1825. doi: 10.1016/j.bbmt.2017.07.021. Epub 2017 Jul 25. PMID 28754544
- [Background] Kutty SS, Peng Q, Danford DA, Fletcher SE, Perry D, Talmon GA, Scott C, Kugler JD, Duncan KF, Quiros-Tejeira RE, Kutty S; Liver Adult-Pediatric-Congenital-Heart-Disease Dysfunction Study (LADS) Group. Increased hepatic stiffness as consequence of high hepatic afterload in the Fontan circulation: a vascular Doppler and elastography study. Hepatology. 2014 Jan;59(1):251-60. doi: 10.1002/hep.26631. Epub 2013 Nov 19. PMID 23913702
- [Background] Dillman JR, Heider A, Bilhartz JL, Smith EA, Keshavarzi N, Rubin JM, Lopez MJ. Ultrasound shear wave speed measurements correlate with liver fibrosis in children. Pediatr Radiol. 2015 Sep;45(10):1480-8. doi: 10.1007/s00247-015-3345-5. Epub 2015 Apr 8. PMID 25851300
- [Background] Karlas T, Weber J, Nehring C, Kronenberger R, Tenckhoff H, Mossner J, Niederwieser D, Troltzsch M, Lange T, Keim V. Value of liver elastography and abdominal ultrasound for detection of complications of allogeneic hemopoietic SCT. Bone Marrow Transplant. 2014 Jun;49(6):806-11. doi: 10.1038/bmt.2014.61. Epub 2014 Apr 7. PMID 24710567
- [Background] Reddivalla N, Robinson AL, Reid KJ, Radhi MA, Dalal J, Opfer EK, Chan SS. Using liver elastography to diagnose sinusoidal obstruction syndrome in pediatric patients undergoing hematopoetic stem cell transplant. Bone Marrow Transplant. 2020 Mar;55(3):523-530. doi: 10.1038/s41409-017-0064-6. Epub 2018 Jan 15. PMID 29335626
- [Background] Barr RG, Ferraioli G, Palmeri ML, Goodman ZD, Garcia-Tsao G, Rubin J, Garra B, Myers RP, Wilson SR, Rubens D, Levine D. Elastography Assessment of Liver Fibrosis: Society of Radiologists in Ultrasound Consensus Conference Statement. Radiology. 2015 Sep;276(3):845-61. doi: 10.1148/radiol.2015150619. Epub 2015 Jun 16. PMID 26079489
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Fontanilla T, Hernando CG, Claros JC, Bautista G, Minaya J, Del Carmen Vega M, Piazza A, Mendez S, Rodriguez C, Aranguena RP. Acoustic radiation force impulse elastography and contrast-enhanced sonography of sinusoidal obstructive syndrome (Veno-occlusive Disease): preliminary results. J Ultrasound Med. 2011 Nov;30(11):1593-8. doi: 10.7863/jum.2011.30.11.1593. PMID 22039033
- [Background] Son CY, Kim SU, Han WK, Choi GH, Park H, Yang SC, Choi JS, Park JY, Kim DY, Ahn SH, Chon CY, Han KH. Normal liver elasticity values using acoustic radiation force impulse imaging: a prospective study in healthy living liver and kidney donors. J Gastroenterol Hepatol. 2012 Jan;27(1):130-6. doi: 10.1111/j.1440-1746.2011.06814.x. PMID 21679249
- See also: D'Souza A ZX. Current Uses and Outcomes of Hematopoietic Cell Transplantation (HCT): CIBMTR Summary Slides, 2016. — https://www.cibmtr.org/ReferenceCenter/SlidesReports/SummarySlides/pages/index.aspx
- See also: Cozadd B (2018) Jazz Pharmaceuticals. 36th Annual JP Morgan Annual Healthcare Conference, San Francisco, California. — https://www.jpmorgan.com/global/healthcareconference
- See also: (2016) In Brief: Defibrotide (Defitelio) for Hepatic Veno-Occlusive Disease. The Medical Letter — https://secure.medicalletter.org/w1503c

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients Enrolled
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients Enrolled
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Between SWE Exams for VOD/SOS
Description: We performed SWE exams once a week for all of our patients. We looked at when patients met clinical criteria for VOD/SOS and then we looked at the SWE exams that were performed before the clinical diagnosis. If the exam immediately preceding the date of clinical diagnosis crossed the threshold for SWE diagnosis, then a frequency of 7 days was sufficient. If it did not, then testing should be more frequent. If multiple preceding exams were positive by SWE, then the optimal testing frequency could be longer than 7 days.
Time Frame: Once a week through study completion assessed for up to 14 weeks
Measure: Mean (Full Range); unit: days
Groups:
- Patients With SOS: Patients who developed SOS during the study period
Arm/Group | Patients With SOS
Number analyzed (Participants) | 6
days | 7 [7 to 7]

2. Secondary Outcome: Determine if SWE Can Provide Earlier SOS Diagnosis Compared to Clinical Criteria.
Description: Number of days where SWE became positive before the clinical criteria became positive.
Time Frame: Daily through study completion assessed for up to 100 days
Measure: Median (Full Range); unit: days
Groups:
- Patients With SOS: Patients who developed SOS during the study
Arm/Group | Patients With SOS
Number analyzed (Participants) | 6
days | 3 [0 to 14]

3. Secondary Outcome: Difference in Maximum SWE Value in Patients With Severe and Very Severe VOD Compared to Those With Mild and Moderate VOD.
Time Frame: Weekly through study completion assessed for up to 14 weeks
Measure: Median (Full Range); unit: percent change from baseline
Groups:
- Patients With Mild/Mod SOS: Patients who developed mild to moderate SOS during the study
- Patients With Severe and Very Severe SOS: Patients who developed severe and very severe SOS during the study
Arm/Group | Patients With Mild/Mod SOS | Patients With Severe and Very Severe SOS
Number analyzed (Participants) | 3 | 3
percent change from baseline | 41 [-2 to 213] | 79 [55 to 91]

4. Secondary Outcome: CEUS Variables Versus Grayscale and Doppler Variables
Description: Quantify relative ability to CEUS parameters versus grayscale and Doppler ultrasound.
  We will compare sensitivity and specificity of time to peak and mean transit time to grayscale and Doppler ultrasound variables for VOD diagnosis.
Time Frame: Study period
Population: Data was not collected for this outcome variables because we can't get the software to collect this data.
Arm/Group | All Patients Enrolled
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | All Patients Enrolled
All-Cause Mortality (participants affected / at risk) | 9/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
Early termination and data necessary for statistical analysis was not collected before research approval expired. The IRB closed the study, requiring the data to since be de-identified. There is no accessible data available to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03858530/Prot_001.pdf
  • Informed Consent Form (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT03858530/ICF_003.pdf